CLINICAL TRIAL: NCT03187782
Title: The Effect of Acupuncture Treatment of Acupoint San Yin Jiao on the Pulse Diagnoses in Patients While Dysmenorrhea is Attacking
Brief Title: Pulse Diagnoses in Patients While Dysmenorrhea is Attacking
Status: Completed | Type: Observational
Sponsor: Taipei Hospital, Taiwan (Other)
Responsible Party: Principal Investigator, Chen-Kai Liao, Doctor, Taipei Hospital, Taiwan
Other Study IDs: TH-IRB-0014-0002
Record Dates: First submitted 2017-05-25; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

INTERVENTIONS:
Diagnostic Test: ANSWatch

SUMMARY:
The mechanism led to the dysmenorrhea can be understood more clearly and one may have a better idea to treat the disease in the future.

DETAILED DESCRIPTION:
Background: Pulse diagnosis of the dysmenorrhea patients before and after acupuncture treatment on the acupoint San Yin Jiao (SP6) were performed so that the mechanism led to the pain can be understood more clearly and one may have a better idea to treat the disease in the future.

Methods: Fifteen women participated in the study voluntarily. They have first to fill in the form of Visual Analogue Scale (VAS) for pain. Then the pulse of the subjects were measured by ANSWatch before and after acupuncture. All meridians can be assessed by analyzing the pulse spectra through Fast Fourier Transform (FFT) of the original pulse data. The significant change of amplitude in certain harmonics which corresponds to a specific meridian after acupuncture treatment can be selected out.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the subjects were the presence of pain during menstruation or three days before it. It needed to recheck if the menstrual cycle appeared within three days after recruiting if dysmenorrhea attacked before menstruation.

Exclusion Criteria:

* The exclusion criterion was that subjects did not take pain killers in the 12 hours before measurement.

Ages: 12 Years to 55 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Fifteen patients suffering from dysmenorrhea who visited the traditional Chinese medicine outpatient department were recruited voluntarily in this study.
  All subjects live in the greater Taipei area.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Patients' radial artery pulses. Change is being assessed. | Measure subjects' radial artery pulses before and after acupuncture in 10 minutes respectively.
  Get subjects' pulses by ANSWatch

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Kai Liao, Principal Investigator — Taipei Hospital

IPD SHARING:
Plan to Share IPD: Undecided